CLINICAL TRIAL: NCT05632913
Title: A Feasibility and Safety Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Recurrent Lung Cancer
Brief Title: Alpha Radiation Emitters Device for the Treatment of Recurrent Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-LUNG -00
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-01

CONDITIONS: Recurrent Lung Cancer; Lung Cancer
Keywords: Alpha radiation; Lung cancer; Recurrent lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seed
  Interventions: Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT)

INTERVENTIONS:
Device: Radiation: Diffusing Alpha Radiation Emitters Therapy (DaRT) — An intratumoral insertion of radioactive sources [Ra-224 containing stainless-steel 316LVM tubes- (Alpha DaRT seeds)]. The seeds release by recoil into the tumor short-lived alpha-emitting atoms

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for treatment of recurrent Lung Cancer .

DETAILED DESCRIPTION:
This is a prospective , interventional, open label, single arm, single center study.

The study is designed to evaluate the Feasibility and Safety of DaRT seeds for the treatment of Recurrent Lung Cancer. The study will be comprised of a screening period, DaRT insertion visit, acute follow-up phase of 4- 8 weeks and a long-term follow up phase of 3 months. The total duration of the study will be 3 months from the DaRT insertion procedure.

A total of 10 subjects will be enrolled to the study .

Eligible patients who meet inclusion/exclusion criteria (as assessed during the screening period) will be invited to the site for the procedure of DaRT seeds insertion. The patients will be monitored for a period of 3 months post insertion

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically proven recurrent mediastinal tumors
* Target lesion is technically amenable for at least 50% coverage by the Alpha DaRT seeds as determined by the treating physician
* Up to two treatable lesions
* Interstitial radiation indication validated by a multidisciplinary team.
* Measurable lesion per RECIST (version 1.1) criteria
* Lesion size ≤ 3 cm in the longest diameter
* Age ≥18 years old
* ECOG Performance Status Scale ≤ 3
* Life expectancy is more than 6 months
* WBC ≥ 3500/µl, granulocyte ≥ 1500/µl
* Platelet count ≥60,000/µl
* Calculated or measured creatinine clearance ≥ 60cc/min. Calculated, or measured creatinine clearance can be≥ 40cc/min given stability of creatinine levels over the past three weeks (at least 1 test per week).
* AST and ALT ≤ 2.5 X ULN
* INR < 1.4 for patients not on Warfarin
* Subjects are willing and able to sign an informed consent form
* Women of childbearing potential (WOCBP) will have evidence of negative pregnancy test before the Ra-224 implantation and are required to use an acceptable contraceptive method to prevent pregnancy for 3 months after brachytherapy.

Exclusion Criteria:

* Concomitant chemotherapy or immunotherapy
* Brain metastases Connective tissue disease (scleroderma, lupus)
* Known hypersensitivity to any of the components of the treatment.
* Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids.
* Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
* Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Patient requires treatment not specified in this protocol which may conflict with the endpoints of this study including evaluation of response or toxicity of DaRT.
* Patients must agree to use adequate contraception (vasectomy or barrier method of birth control) prior to study entry, for the duration of study participation and for 3 months after discontinuing therapy.
* Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of DaRT.
* High probability of protocol non-compliance (in opinion of investigator).
* Breastfeeding women or women of childbearing potential unwilling or unable to use an acceptable contraceptive method to prevent pregnancy for 3 months after RT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility - DaRT seed placement | From Day 0-Day 90
  Feasibility will be determined according to the rate of successful placement of DaRT seeds via imaging
Safety- Adverse events | From Day 0-Day 90
  Safety will be determined according to the overall incidence of device related SAE's graded according to CTCAE v5.0 criteria

SECONDARY OUTCOMES:
Efficacy - Alpha DaRT seeds | 1 month and 3 months
  Local control evaluation according to RECIST v1.1
Efficacy - Alpha DaRT seeds | Day 0-Day 90
  Tumor Coverage

CONTACTS AND LOCATIONS:
Overall Officials: Aron Popovtzer, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah University Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No